CLINICAL TRIAL: NCT01211249
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter, Exploratory Phase II Study to Compare Three Dose Regimens of GLPG0259 vs Placebo, in Combination With Methotrexate, Administered for 12 Weeks to Subjects With Active Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Brief Title: GLPG0259 in Methotrexate-refractory Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0259-CL-201; 2009-015898-12 (EudraCT Number)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate-refractory
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GLPG0259 (Part A) (Experimental)
  Interventions: Drug: GLPG0259 oral capsule
- Placebo (Part A) (Placebo Comparator)
  Interventions: Drug: Placebo
- GLPG0259 (Part B) (Experimental)
  Interventions: Drug: GLPG0259 (Part B)
- Placebo (Part B) (Placebo Comparator)
  Interventions: Drug: Placebo (Part B)

INTERVENTIONS:
Drug: GLPG0259 oral capsule — Two capsules, each containing 25 mg of GLPG0259 (i.e. 50 mg/day), to be given once daily; in case of adverse events the dose may be split over two administrations, or reduced to 25 mg/day (one single capsule)
  Arms: GLPG0259 (Part A)
Drug: Placebo — Placebo capsules; two capsules to be taken in the morning, in case of adverse events the dose may be split over two administrations, or reduced to one single capsule
  Arms: Placebo (Part A)
Drug: GLPG0259 (Part B) — Capsule, dosage to be established based on results of Part A
  Arms: GLPG0259 (Part B)
Drug: Placebo (Part B) — Capsules, dosage to be established after Part A, and matching GLPG0259 (Part B)
  Arms: Placebo (Part B)

SUMMARY:
Part A: 30 patients suffering from active rheumatoid arthritis despite continued treatment with methotrexate will receive once daily two capsules containing either GLPG0259 (25 mg/capsule) or matching placebo, for 12 weeks. In the course of the study the patients will be examined for severity of disease, as well as for any adverse effects that may occur. If needed, dosing may be split to one capsule twice daily, or reduced to one capsule of 25 mg.

Part B: If results of Part A suggest test medication to have a therapeutic advantage over placebo and to be well-tolerated, more patients will be recruited for Part B, where various dosages will be assessed. These dosages will be established based on results from Part A.

ELIGIBILITY:
Inclusion Criteria:

* Must have active RA (≥5 tender or painful joints on motion and ≥5 joints swollen AND a C-reactive protein (CRP) concentration ≥1.5 mg/dL).
* Must have been on methotrexate for ≥6 months at a stable dose of 7.5-25 mg/week for ≥12 weeks, to be continued throughout study;
* If on oral steroids, these should be at a dose ≤10 mg/day of prednisone eq and stable for ≥4 weeks prior to screening;
* If on NSAIDs, these must be at a stable dose for ≥2 weeks prior to screening;
* Women must have negative pregnancy test unless surgically sterile or post-menopausal for ≥1 year;
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for ≥12 weeks after the last dose of study drug.
* Informed consent

Exclusion Criteria:

* Must not have received treatment with DMARDs, other than background methotrexate;
* Must not be receiving or have received RA treatment with a biological agent, except if administered in a clinical study ≥six months prior to screening (12 months for rituximab or other B cell depleting agents);
* Must not have received any treatment with a cytotoxic agent, other than methotrexate, before screening (e.g. chlorambucil, cyclophosphamide, nitrogen mustard, or other alkylating agents);
* Must not have received intra-articular or parenteral corticosteroid injection within four weeks prior to screening;
* Must not regularly be using aspirin or any other anti-coagulant medication;
* Must not have a known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the Investigator, such as anaphylaxis, requiring hospitalization;
* Must not have positive serology for human immunodeficiency virus (HIV)1 or 2 or hepatitis B or C, or any history of HIV or hepatitis from any cause with the exception of hepatitis A;
* Must not have a history of any inflammatory rheumatological disorders other than RA;
* Must not have undergone (or planned) surgical treatments for RA;
* Must not have symptoms of clinically significant illness other than RA (including but not limited to cardiopulmonary, renal, metabolic, hematologic, or psychiatric disorders) within three months prior to screening;
* Must not have a history of active infections requiring intravenous antibiotics within the past four weeks;
* Must not have a history of malignancy within the past five years (except for basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been treated with no evidence of recurrence);
* Must not have a history of tuberculosis (TB) infection as determined by a positive diagnostic TB test result (defined as a positive QuantiFERON TB Gold test), AND a recent chest radiograph (both posterior-anterior and lateral views), read by a qualified radiologist, with evidence of current active TB or old inactive TB.
* Must not have been administered a live vaccine within four weeks prior to screening;
* Must not have participated in any investigational drug/device clinical study within four weeks prior to screening, in biological agents clinical studies within six months prior to screening, and B cell-depleting agent clinical studies within 12 months prior to screening;
* Must not have a history within the previous two years or current evidence of drug or alcohol abuse;
* Must not have any condition or circumstances which in the opinion of the Investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements, or may pose a risk to the patient's safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 weeks
  The primary efficacy endpoint will be the number and percentage of subjects in each GLPG0259 dose group and placebo group achieving an American College of Rheumatology (ACR)20 (ACR20 response rate) at Week 12.

SECONDARY OUTCOMES:
Efficacy | intermediate timepoints for 12 weeks
  ACR20, ACR50, ACR75 and DAS28 (and components) at weeks 1, 2, 4, 8 and 12;
Safety | 12 weeks
  At each return visit, patients will be asked about adverse events, and undergo examination of heart (ECG) and bloodpressure; blood- and urine-samples will be collected to monitor organ functions.
Pharmacokinetics | 12 weeks
  On several timepoints throughout the study bloodsamples will be taken from the patient to establish the amount of the study medication in the blood, and to determine how long it stays in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PhD, Study Director — Galapagos NV
Locations (32):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - KU Leuven, Leuven
  - AZ Alma, Sijsele-Damme
- UMC Leiden, Leiden, Netherlands
- Poland (5):
  - Specjalistyczne Centrum Medyczne NZOZ NOWOMED, Krakow
  - "Linea Corporis" - Chirurgia Plastyczna Sp. z o.o., Warsaw
  - Mokotowskie Centrum Osteoporozy S.C., Warsaw
  - Synexus SCM Sp. z o.o., Wroclaw
  - Akademia Medyczna im. Piastów Śląskich we Wroclawiu Katedra i Klinika Reumatologii i Chorób Wewnętrznych UM we Wrocławiu, Wroclaw
- Russia (13):
  - State Educational Institution of Higher Professional Education "Moscow State Medico-Stomatological University of Roszdrav" State Healthcare Institution of City Moscow "City Clinical Ordena Trudovogo Krasnogo Znameny Hospital #23 n.a. "Medsantrud", Moscow
  - State Healthcare Institution of city Moscow "City Clinical Ordena Trudovogo Krasnogo Znameny Hospital #23 n.a. "Medsantrud", Moscow
  - State Educational Institution of Higher Professional Education "Russian State Medical University of Roszdrav" State Healthcare Institution of City Moscow "City Clinical Hospital #15 n.a. O.M. Filatov", Moscow
  - State Healthcare Institution of City Moscow "City Clinical Hospital #4", Moscow
  - State Healthcare Institution of City Moscow "City Clinical Hospital #7", Moscow
  - Institution Russian Academy of Medical Sciences Scientific Research Institution of Rheumatology RAMN, Moscow
  - State Healthcare Institution of City Moscow "City Clinical Hospital #1 n.a. Pirogov", Moscow
  - State Educational Institution of Higher Professional Education "Moscow State Medico-Stomatological University of Roszdrav" at the State Healthcare Institution of city Moscow "City Clinical Ordena Trudovogo Krasnogo Znameny hospital #23 n.a. "M, Moscow
  - Saint-Petersburg State Healthcare Institution "City Hospital #26", Moscow
  - Saint-Petersburg State Healthcare Institution "City Pokrovskaya Hospital", Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "City Mariinskiy Hospital", Saint Petersburg
  - Institution of Russian Academy of Sciences Saint-Petersburg Clinical Hospital RAN, Saint Petersburg
  - State Educational Institution of Higher Professional Education "Saint-Petersburg State Pediatric Medical Academy of Roszdrav", Saint Petersburg
- Ukraine (10):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Donetsk City Hospital No5, Donetsk
  - Kharkiv City Clinical Hospital No.27, Kharkiv
  - Kharkiv City Clinical Hospital No.8, Kharkiv
  - Kyiv City Clinical Hospital No.3, Kyiv
  - Central Pool-type Clinical Hospital MoH of Ukraine, Kyiv
  - Institute of Gerontology AMS of Ukraine, Kyiv
  - University Clinic, Crimean Medical University, Simferopol
  - Vinnytsia Regional Hospital, Vinnytsia
  - Zaporizhzhia Regional Hospital, Zaporizhzhya

REFERENCES:
- [Derived] Westhovens R, Keyser FD, Rekalov D, Nasonov EL, Beetens J, Van der Aa A, Wigerinck P, Namour F, Vanhoutte F, Durez P. Oral administration of GLPG0259, an inhibitor of MAPKAPK5, a new target for the treatment of rheumatoid arthritis: a phase II, randomised, double-blind, placebo-controlled, multicentre trial. Ann Rheum Dis. 2013 May;72(5):741-4. doi: 10.1136/annrheumdis-2012-202221. Epub 2012 Nov 17. PMID 23161899